CLINICAL TRIAL: NCT03788148
Title: Bare-metal Stents(BMS) Versus Drug-eluting Stents(DES) in Patients Who Underwent Periprocedural Blood Transfusion : A Nationwide Longitudinal Cohort Study
Brief Title: Bare Metal Stents and Drug Eluting Stents in Patients Who Underwent Blood Transfusion
Acronym: TFPCI2
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Ho Choi, MD, PhD, Professor, Principal Investigator, Samsung Medical Center
Other Study IDs: SMC 2017-11-132
Record Dates: First submitted 2018-12-14; First posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Erythrocyte Transfusion; Percutaneous Coronary Intervention; Revascularization
Keywords: transfusion, PCI, DES, BMS
MeSH Terms: conditions — Dysequilibrium syndrome | interventions — Stents; Erythrocyte Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stent, red blood cell transfusion — BMS (Bare Metal Stent) and DES (drug-eluting stent) transplants with periprocedural red blood cell transfusion

SUMMARY:
Retrospective cohort study of Korean National Healthcare Insurance Database. To investigate clinical outcomes of bare metal stents versus drug eluting stents in patients who underwent periprocedural red blood cell transfusion.

DETAILED DESCRIPTION:
A Korean nationwide, multi-center, retrospective observational cohort study.

The receipt of red blood cell transfusion is at high risk of cardiac events or death. But little is know regarding the comparative outcomes of BMS and DES implantation in patients who underwent periprocedural red blood cell transfusion.

Longitudinal data is collected from administrative claims in the national health insurance services of Korea. All Korean data(N=500,591) undergoing PCI from 2006 to 2015 is extracted. BMS or DES Patients(N=28,322) who received periprocedural red blood cell transfusion is investigate. Clinical outcomes until December 31, 2017 is investigate.

Primary endpoint is a time to the first major adverse clinical event(MACE) defined as a composite of all-cause death, revascularization, critically ill cardiovascular status, or stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with percutaneous coronary intervention from 2006 to 2015
* Patients with the implantation of BMS or DES
* Patients with the receipt of periprocedural red blood cell transfusion

Exclusion Criteria:

* Patients without any of stent implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Korean patients undergoing BMS or DES implantation from January 1, 2005 to December 31, 2016 who received periprocedural red blood cell transfusion
Sampling Method: Non-Probability Sample
Enrollment: 28322 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence density of MACE (Major adverse clinical events) | 3 years
  The first major adverse clinical event(MACE) defined as a composite of all-cause death, revascularization, critically ill cardiovascular status, and stroke.
Incidence density of MACE (Major adverse clinical events) | 1 year
  The first major adverse clinical event(MACE) defined as a composite of all-cause death, revascularization, critically ill cardiovascular status, and stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ho Choi, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gang nam-Gu, Ilwon-Dong, South Korea

IPD SHARING:
Plan to Share IPD: No